CLINICAL TRIAL: NCT06997575
Title: Frequency of Recurrence of Seizures With Intravenous Versus Intramuscular Magnesium Sulphate in Women With Eclampsia
Brief Title: Comparing Intravenous and Intramuscular Magnesium Sulphate for Preventing Seizure Recurrence in Women With Eclampsia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nishtar Medical University (Other)
Responsible Party: Principal Investigator, Dr. Laraib Irshad, Principal Investigator, Nishtar Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1323-1123
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Eclampsia; Seizures; Pregnancy
Keywords: Magnesium sulphate; eclampsia; Seizures; intramuscular; intravenous
MeSH Terms: conditions — Eclampsia; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Patients will receive 4 g of Intravenous MgSO4 as 20% solution followed by 1 g Intravenous per hour as continuous IV infusion. MgSo4 will be continued for 24 h after the last seizure or 24 h after delivery, whichever will occur last.
  Interventions: Drug: Magnesium Sulphate infusion
- Group B (Experimental): Patients initially will receive a 10 g loading dose of MgSO4: 4 g will be given Intravenous as 20% solution, 6 g IM 50% solution divided equally 3 g in each buttock with 1% of 1 ml of lidocaine) followed by 2.5 g IM every 4 h as maintenance therapy. MgSo4 will be continued for 24 h after the last seizure or 24 h after delivery, whichever will occur last.
  Interventions: Drug: Magnesium Sulphate infusion; Drug: Magnesium sulphate intramuscular

INTERVENTIONS:
Drug: Magnesium Sulphate infusion — Infusion of 20% MgSO4 solution
  Other Names: magnesium sulphate intravenous
Drug: Magnesium sulphate intramuscular — Intramuscular injections will be instituted in gluteal region.
  Other Names: MgSO4 intramuscular
  Arms: Group B

SUMMARY:
The goal of this clinical study is to learn whether the way we give magnesium sulphate-into a vein (intravenous, IV) versus into a muscle (intramuscular, IM)-affects how often women with eclampsia have repeat seizures.

The main question it aims to answer is:

1. Do women who receive IV magnesium sulphate have fewer recurrent seizures than those who receive IM magnesium sulphate?

Researchers will compare two groups of women with eclampsia: one group will receive a bolus and a continuous IV infusion of magnesium sulphate, and the other will receive a combined IV-plus-IM dosing regimen.

Participants will:

1. Be women aged 18-45 years diagnosed with eclampsia in the labour room.
2. Have their basic health information (age, gestation, parity, body mass index) recorded
3. Be randomly assigned (by sealed envelope) to receive either the IV regimen (4 g loading dose then 1 g/hour infusion) or the IM regimen (10 g loading dose with 4 g IV plus 6 g IM, then 2.5 g IM every 4 hours).
4. Continue treatment for 24 hours after their last seizure or delivery, whichever is later.
5. Be monitored in hospital for seizure recurrence.
6. Have any repeat seizure treated immediately with an extra IV dose of magnesium sulphate.

ELIGIBILITY:
Inclusion Criteria:

* Admitted in labor room due to eclampsia (new onset of grand mal seizure activity and/or unexplained coma during pregnancy)

Exclusion Criteria:

* Patients with intracranial bleeding (on CT-scan)
* Already received MgSO4, phenytoin and diazepam before attending the hospital

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women with eclampsia
Enrollment: 200 (Actual)
Dates: Start 2025-05-13 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Seizure | Within 48 hours after the last dose of MgSO4
  Seizure recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Mehnaz Khakwani Professor, FCPS, Study Chair — Nishtar Medical University & Hospital Multan
Locations (1):
- Nishtar Medical University & Hospital, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saha PK, Kaur J, Goel P, Kataria S, Tandon R, Saha L. Safety and efficacy of low dose intramuscular magnesium sulphate (MgSO4) compared to intravenous regimen for treatment of eclampsia. J Obstet Gynaecol Res. 2017 Oct;43(10):1543-1549. doi: 10.1111/jog.13424. Epub 2017 Jul 16. PMID 28714170